CLINICAL TRIAL: NCT01892241
Title: Efficacy and Safety of Peginterferon a-2a in Patients of Chronic Hepatitis B With Spontaneous Decline of HBV DNA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Cai Qingxian, Doctor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATFSHBVD
Record Dates: First submitted 2012-08-22; First posted 2013-07-04 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Antiviral Treatment of Chronic Hepatitis B
Keywords: Chronic hepatitis B,Spontaneous Decline of HBV DNA,Peginterferon a-2a, entecavir
MeSH Terms: interventions — peginterferon alfa-2a; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 180µg of peginterferon alfa-2a (Experimental): Cases in group A receive 180µg of peginterferon alfa-2a (Pegasys,Roche) once weekly for 48 weeks.
  Interventions: Drug: Pegasys(Roche)
- Entecavir (Active Comparator): cases in group B received an continual entecavir therapy(0.5 mg orally once daily)
  Interventions: Drug: Entecavir
- Control group (No Intervention): Those in group C didn't accept any antiviral regiment .

INTERVENTIONS:
Drug: Pegasys(Roche) — 180µg of peginterferon alfa-2a (Pegasys,Roche) once weekly for 48 weeks.
  Other Names: peginterferon alfa-2a
  Arms: 180µg of peginterferon alfa-2a
Drug: Entecavir — continual entecavir therapy(0.5 mg orally once daily)
  Arms: Entecavir

SUMMARY:
Patients with spontaneous decline of HBV DNA were non-randomly assigned to accept peginterferon alfa-2a or entecavir therapy, or didn't accept any antiviral regiment.

DETAILED DESCRIPTION:
It was a prospective, non-randomized, open-label study that evaluated the efficacy and safety of pegasys treatment in chronic hepatitis B patients with spontaneous HBVDNA decline after acute exacerbation.Patients with spontaneous decline of HBV DNA(a decrease of HBV DNA levels of more than 2 log(10) IU/mL as compared to baseline before antiviral treatment) after acute exacerbation (ALT was 10-30ULN，TBIL was 2-20mg/ml，PTA>60%)were non-randomly divided into 3 groups: group A, B and C. Before treatment, the patients were counselled on the advantages and disadvantages of taking peginterferon or nucleos(t)ide analogue, and the subsequential treatment were decided by themselves. Cases in group A receive 180µg of peginterferon alfa-2a (Pegasys,Roche) once weekly for 48 weeks. Group B and C were control group, cases in group B received an continual entecavir therapy(0.5 mg orally once daily) and those in group C didn't accept any antiviral regiment.

ELIGIBILITY:
This study focused on the subsequential antiviral therapeutic strategies for chronic hepatitis B patients with spontaneous decline of HBV DNA after acute exacerbation. Patients fullfilled the following criterias were chosen for screening: They were antiviral treatment naı¨ve and had been positive for hepatitis B surface antigen (HBsAg) for at least 6 months, were positive for HBeAg and had an HBV DNA Level of more than 500,000IU/ml. Their serum alanine aminotransferase level was greater than 2 but less than or equal to 30 times the upper limit of the normal range, their peak value of total bililubin ranged from 2mg/ml to 20mg/ml and the prothrombin time activity was greater than 60%.

ALL of these patients were hospitalized and pretreated with anti-inflammation and liver protection agents such as Stronger Neo-Minophagen C, Polyunsaturated phosphatidylcholine (Essentiale), Ursodeoxycholic Acid and L-Glutathione reduced, without any nuclutide of nucleoside. Their ALT、TBIL and PTA were monitor weekly and HBVDNA level were measured every two weeks. Patients were eligible if their HBVDNA declined spontaneously by 2 log(10) IU/mL while their ALT falled below 10 ULN and TBIL falled below 2mg/ml within 8 weeks of pretreatment.

Patients with advanced fibrosis, cirrhosis and hepatoma were excluded. Other cause of chronic liver disease should be systematically checked to exclude co-infection with HDV, HCV and HIV, comorbidities with alcoholism, autoimmune and metabolic liver disease. Serious medical or psychiatric illnesses that had usage of corticosteroid or immunosup-pressive agents at the time of study were excluded. All patients in this study lived in Guangdong, a province of 100,000,000 populations, with same demographics. Owing to patients fear or refusal of liver biopsy, no patients had the liver biopsy and the rest relied on other clinical methods to obtain equivalent information of patient conditions. In our cases, ultrasonorgraphy helped to filter out patients with advanced fibrosis.The liver sonar examination was performed by two experi-enced hepatologists at least three times on each patient.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Complete viralogic response | week 96
  Complete viralogic response was defined as suppression of HBV DNA to the level below 60IU/mL(detected by Cobas Amplicor HBV Monitor Test, Roche Diagnostics).

SECONDARY OUTCOMES:
HBsAg loss and seroconversion | week 24,48,72 and 96
  HBsAg loss was defined as HBsAg titre less than 0.05 IU/mL and the HBsAg seroconversion was defined as the loss of HBsAg and the presence of anti-HBs antibody. HBeAg seroconversion was defined as disappearance of HBeAg and appearance of anti-HBe antibody, while HBeAg loss was defined as disappearance of HBeAg only.
ALT normalization | week 24,48,72 and 96
  ALT normalization was defined as ALT level less than 40 IU/L(determined by a sequential multiple autoanalyzer).
Sick leave in patients in different groups | week 48,72 and 96

CONTACTS AND LOCATIONS:
Overall Officials: Gao Zhiliang, doctor, Study Chair — The Third Affliated Hospital of Sun Yat-sen University; Zhao Zhixin, doctor, Study Director — The Third Affliated Hospital of Sun Yat-sen University